CLINICAL TRIAL: NCT05231421
Title: A Focus Group Study to Explore Smoking Triggers and Acceptability of Just-in-time Adaptive Interventions (JITAI) for Smoking Cessation Among Low-income Smokers
Brief Title: A Focus Group Study to Explore Smoking Triggers and Acceptability of Just-in-time Adaptive Intervent
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 19-2555.cc
Record Dates: First submitted 2021-12-21; First posted 2022-02-09 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Smoking; Smoking Cessation; Smoking Behaviors
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Low-income smokers: Interested participants will first complete a screening survey asking about their demographic information and checking whether are eligible for this study. If eligible, participants will read a consent statement. Only those who give consent would be allowed to proceed. If participants agree to be in this study, they will continue to participate in the study and schedule a time for focus group discussion.
  Interventions: Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Focus Group — Each focus group will consist of 5-10 participants. They will first introduce to each other and be asked to keep information shared during the session private. The moderator will initiate some questions for the group to discuss. Prompt and follow-up questions will be asked. There is no right or wrong answer for each question and no sensitive questions will be asked. The conversations during the focus group discussion will be recorded. The group will be debriefed about the purpose of the study and have a chance to ask any questions about the study if they have. The focus group discussion for each session will last about 60-90 minutes.

SUMMARY:
This research intends to identify common smoking triggers and barriers to quitting smoking; understand useful and effective strategies for smoking cessation; and explore the feasibility and acceptability of mobile phone-based interventions among low-income smokers.

DETAILED DESCRIPTION:
This research intends to identify common smoking triggers and barriers to quitting smoking; understand useful and effective strategies for smoking cessation; and explore the feasibility and acceptability of mobile phone-based interventions among low-income smokers.

Specific research questions of this research project are:

1. What are the common smoking triggers and barriers to quitting smoking for low-income smokers?
2. What are the preferred and useful smoking cessation strategies based on low-income smokers quitting experience?
3. What is the feasibility and acceptability of using a) text messages, b) virtual reality programs, and c) just-in-time adaptive smoking cessation interventions among low-income smokers?

ELIGIBILITY:
Inclusion criteria:

1. between 18 and 89 years old
2. current smokers
3. reside in Denver Metropolitan Area
4. have a personal cell phone
5. have a household income at or lower than 200% of the federal poverty level; and
6. ability to read and speak English or Spanish (since a large proportion of the low-SES population in Denver are Spanish speakers).

Exclusion criteria:

1. Unable to provide informed consent;
2. age ≥ 89 years;
3. unable to speak or understand English, or Spanish.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit low-income current smokers
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Use focus group discussion to identify barriers faced by low-income smokers | 12 months
  This study intends to identify the barriers faced by low-income smokers to obtaining smoking cessation services/support using focus groups of current smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Zhou, Principal Investigator — Colorado Research Center
Locations (1):
- Colorado Research Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No